CLINICAL TRIAL: NCT04072471
Title: Post-Authorisation Safety Study of Lesinurad
Acronym: SATURATES
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn as lesinurad was withdrawn from the market in Europe by the market authorization holder. Hence the commitment to do this PASS was removed by the European Medicines Agency.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5310R00016; EUPAS30385 (Registry Identifier: EU PASS Register)
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — lesinurad

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zurampic®: Patients exposed to Zurampic® plus a xanthine oxidase inhibitor (allopurinol or febuxostat) (lesinurad+XOI)
  Interventions: Drug: Zurampic®
- Control group: xanthine oxidase inhibitor monotherapy: Patients exposed to xanthine oxidase inhibitor monotherapy (allopurinol or febuxostat).
  Interventions: Drug: Control group: xanthine oxidase inhibitor monotherapy

INTERVENTIONS:
Drug: Zurampic® — non-interventional study where patients are exposed to Zurampic® plus a xanthine oxidase inhibitor (allopurinol or febuxostat) during the normal course of clinical practice
  Other Names: ATC code: M04A B05; Product name*: Zurampic®; Substance (INN)*: lesinurad
  Groups: Zurampic®
Drug: Control group: xanthine oxidase inhibitor monotherapy — non-interventional study where patients are exposed to xanthine oxidase inhibitor monotherapy (allopurinol or febuxostat) during the normal course of clinical practice
  Groups: Control group: xanthine oxidase inhibitor monotherapy

SUMMARY:
Non-interventional population-based prospective cohort study in multiple databases comparing patients with gout who initiate lesinurad in combination with an existing xanthine oxidase inhibitor (XOI) (lesinurad+XOI cohort) to a propensity score-matched cohort of similar patients from the same data source who continue treatment with XOI monotherapy (XOI mono cohort). Study will characterize the cardiovascular safety of lesinurad in combination with XOI in patients with gout aged 18+ years compared with similar patients who continue XOI monotherapy. Primary objective: to assess the relative incidence of major adverse cardiac events plus hospitalization for unstable angina (MACE+ events) in patients with gout in both cohorts. Secondary objectives: to describe the characteristics of the cohorts prior to matching; to assess the relative incidence of hospitalisation for acute kidney injury between the matched cohorts; to assess the relative incidence of individual MACE+ components in the matched cohorts.

ELIGIBILITY:
Inclusion Criteria:

* More than one dispensing/prescription for an xanthine oxidase inhibotor (XOI) within the past 183 days prior to the index date and days' supply extending beyond the index date
* A coded diagnosis of gout at any time in the past or on the index date
* Age 18 years or older
* Continuous enrolment in the database for the past 183 days

Exclusion Criteria:

* Patients on urate-lowering therapy medications within 6 months prior to the index date to manage gout (probenecid, benzbromarone, or pegloticase) other than an XOI (allopurinol, febuxostat) or lesinurad (not including medications to treat gout flares).
* Patients with severe renal impairment defined using clinical diagnostic codes (i.e., a diagnosis code of CKD stage IV, end-stage renal disease, or an indicator that eCrCl is < 30 mL/min at any time prior to the index date).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in this study will be 18 years of age or older, will have had at least 6 months (183 days) of continuous baseline data available before entering one of the cohorts, and will be current users of XOI monotherapy (i.e., > 1 dispensing/prescription of a study XOI in the 183-day baseline period prior to the index date and days' supply extending beyond the index date). The study population will include patients from one primary care database in Italy (Health Search) and another in Spain (Information System for Research in Primary Care [SIDIAP]), as well as two US health systems (the HealthCore Integrated Research DatabaseSM [HIRD] and Medicare).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-29 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE+) | 2 year follow-up
  MACE+ is a composite endpoint comprised of: hospitalisation for non-fatal AMI, stroke, or unstable angina and cardiovascular (CV) death. CV death includes the following causes, occurring in or out of the hospital: AMI, sudden cardiac, heart failure, CV procedures, CV haemorrhage, stroke, underlying cerebrovascular cause, other CV causes.

SECONDARY OUTCOMES:
Hospitalisation for acute kidney injury (AKI) including renal failure (with AKI as the primary diagnosis) | 2 year follow-up
  Confirmed cases of AKI require all three of the following criteria:
  * A diagnosis of renal injury or acute renal injury recorded as a primary hospital discharge diagnosis in the electronic database AND
  * An increase in serum creatinine at hospital admission or within 48 hours of hospital admission defined as follows:
    * Increase in serum creatinine by ≥ 1.5-fold from baseline where baseline is lowest value recorded within 1 year before the hospital admission date OR
    * Decrease in estimated glomerular filtration rate (eGFR) or actual 24-hour GFR by ≥ 50% from baseline where baseline is highest value recorded within 1 year before the hospital admission date OR
    * Estimated creatinine clearance (eCrCl) < 30 mL/min AND
  * Absence of all the following contraindications for lesinurad patients at any time prior to the index date:
    * A diagnosis code of chronic kidney disease stage IV or greater
    * eCrCl < 30 mL/min recorded at any time prior to the index date
Each individual component of MACE+ | 2 year follow-up
  This can be the hospitalisation for non-fatal AMI, stroke, or unstable angina and cardiovascular (CV) death.